CLINICAL TRIAL: NCT03725943
Title: Assessment of the Performance of the V2 Version of the Dreem Headband for EEG Sleep Monitoring Compared to a Gold Standard Polysomnography.
Brief Title: Comparison of Dreem to Clinical PSG for Sleep Monitoring in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dreem (Industry)
Collaborators: Institut de Recherche Biomedicale des Armees (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OCTAVE IRBA
Record Dates: First submitted 2018-10-29; First posted 2018-10-31 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Sleep
Keywords: Automated Sleep Staging

STUDY DESIGN:
Intervention Model Description: Dreem
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy adults (Experimental): Dreem
  Interventions: Diagnostic Test: Dreem

INTERVENTIONS:
Diagnostic Test: Dreem — Dreem Band to be worn by each participant while undergoing in-lab sleep study with PSG.

SUMMARY:
This study aims to evaluate the accuracy of automated sleep analysis by the Dreem dry-EEG headband and deep learning algorithm in comparison to the consensus of 5 sleep technologists' manual scoring of a gold-standard clinical polysomnogram (PSG) record in healthy adult volunteers during an overnight clinic-based sleep study.

DETAILED DESCRIPTION:
The study will enroll 25 adult volunteers who will undergo a one-night in-lab sleep study. All volunteers are first prescreened over the phone. Upon arrival at the research center, volunteers provide informed consent, are interviewed to confirm eligibility, and complete a detailed demographic, medical, health, sleep, and lifestyle survey. After the survey, participants are fitted with the PSG and the Dreem headband by the sleep technologist. During the PSG sleep study, the Dreem headband records EEG, pulse, oxygen saturation (SO2), movement, and respiratory rate.

Dreem's algorithms will be used to automatically stage the Dreem sleep data, and the results will then be compared to the consensus of 5 sleep technologists' manual scoring of the respective PSG records for the same individuals to determine the accuracy of Dreem's sleep staging algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Capable of providing informed consent

Exclusion Criteria:

* Pregnant or nursing females
* History of any severe comorbidities such as cardiac, neurologic, or psychiatric diseases/disorders in the last 12 months
* Morbid obesity (BMI >= 40)
* Use of benzodiazepines, nonbenzodiazepine (Z-drugs), or Gammahydroxybutyrate (GHB) the day/night of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Sleep stages accuracy (Dreem vs. PSG consensus) | Day 1
  Cohen's kappa comparing the classification of AASM sleep stages at each 30-sec epoch determined automatically by the Dreem headband compared those determined by the consensus of 5 sleep technologists' scoring of each subject's PSG record from the same night.

SECONDARY OUTCOMES:
Total Sleep Time (TST) (accuracy between Dreem and PSG consensus) | Day 1
  Total time (in minutes) the subject spends asleep as automatically determined by the Dreem headband compared to the TST determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.
Wake After Sleep Onset (WASO) time (accuracy between Dreem and PSG consensus) | Day 1
  Total time (in minutes) the subject spends awake from sleep onset to sleep end as automatically determined by the Dreem headband compared to the WASO determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.
Time in N1 sleep stage (accuracy between Dreem and PSG consensus) | Day 1
  Total time (in minutes) the subject spends in AASM N1 sleep stage as automatically determined by the Dreem headband compared to the N1 time determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.
Time in N2 sleep stage (accuracy between Dreem and PSG consensus) | Day 1
  Total time (in minutes) the subject spends in AASM N2 sleep stage as automatically determined by the Dreem headband compared to the N2 time determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.
Time in N3 sleep stage (accuracy between Dreem and PSG consensus) | Day 1
  Total time (in minutes) the subject spends in AASM N3 sleep stage as automatically determined by the Dreem headband compared to the N3 time determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.
Time in rapid eye movement (REM) sleep stage (accuracy between Dreem and PSG consensus) | Day 1
  Total time (in minutes) the subject spends in AASM REM sleep stage as automatically determined by the Dreem headband compared to the REM time determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.
Number of sleep slow oscillations (accuracy between Dreem and PSG consensus) | Day 1
  Number of sleep slow oscillations counted automatically by the Dreem headband compared to those determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.
Number of sleep spindles (accuracy between Dreem and PSG consensus) | Day 1
  Number of sleep spindles counted automatically by the Dreem headband compared to those determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.
Number of sleep eye movements (accuracy between Dreem and PSG consensus) | Day 1
  Number of eye movements during sleep counted automatically by the Dreem headband compared to those determined by the consensus of 5 sleep technologists' scoring of the subject's PSG record from the same night.
Breathing frequency measurement (accuracy between Dreem and PSG consensus) | Day 1
  Breathing frequency measured automatically by the Dreem headband's accelerometer compared to those determined by the nasal cannula on the subject's PSG from the same night.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Sauvet, M.D., Ph.D., Principal Investigator — Institut de Recherche Biomédicale des Armées
Locations (1):
- Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge, D19, France

IPD SHARING:
Plan to Share IPD: Undecided
We plan to share de-identified physiological data in an open-source format to the public. However, this will only occur if the data files are of sufficient quality and likely to be of use to the scientific community. This decision may also depend on certain legal or business constraints.

REFERENCES:
- [Derived] Arnal PJ, Thorey V, Debellemaniere E, Ballard ME, Bou Hernandez A, Guillot A, Jourde H, Harris M, Guillard M, Van Beers P, Chennaoui M, Sauvet F. The Dreem Headband compared to polysomnography for electroencephalographic signal acquisition and sleep staging. Sleep. 2020 Nov 12;43(11):zsaa097. doi: 10.1093/sleep/zsaa097. PMID 32433768